CLINICAL TRIAL: NCT04674774
Title: Efficacy of Tegoprazan Based Bismuth Quadruple Therapy Compared With Bismuth Quadruple Therapy for Helicobacter Pylori Infection: Randomized, Double-blind, Active-Controlled Study
Brief Title: Efficacy of Tegoprazan Based Bismuth Quadruple Therapy for Helicobacter Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Incheon St.Mary's Hospital (Other)
Responsible Party: Principal Investigator, Joon Sung Kim, Assistant Professor, Incheon St.Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OC20MIDI0057
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — tegoprazan; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tegoprazan based bismuth quadruple therapy group (Experimental): tegoprazan based bismuth quadruple therapy group
  Interventions: Drug: Tegoprazan
- PPI based bismuth quadruple therapy group (Active Comparator): PPI based bismuth quadruple therapy group
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Tegoprazan — oral administration of tegoprazan-based bismuth quadruple therapy(tegoprazan 50 mg b.i.d, bismuth 300 mg q.i.d, metronidazole 500 mg t.i.d, tetracycline 500 mg q.i.d) for 14 days
  Arms: tegoprazan based bismuth quadruple therapy group
Drug: Lansoprazole — oral administration of PPI-based bismuth quadruple therapy(lansoprazole 30 mg b.i.d, bismuth 300 mg q.i.d, metronidazole 500 mg t.i.d, tetracycline 500 mg q.i.d) for 14 day
  Arms: PPI based bismuth quadruple therapy group

SUMMARY:
This study aims to investigate eradication rate, drug compliance, and adverse events in patients with confirmed Helicobacter pylori infection between tegoprazan, bismuth, metronidazole, and tetracycline for 14 days (TBMT) and PPI, bismuth, metronidazole, and tetracycline for 14 days (LBMT)

DETAILED DESCRIPTION:
This is a multi-center, double-blind, randomized, active-controlled study.

ELIGIBILITY:
Inclusion Criteria:

patients who male or female aged 19 to 75 years old and fall under the following conditions with confirmed helicobacter pylori infection

Exclusion Criteria:

1. patients who have H.pylori eradication history
2. patients with history of gastric cancer surgery
3. patients who have taken antibiotics within 4 weeks prior to trial
4. a person who taking HIV protease inhibitors (atazanavir, nelfinavir) or a drug containing rilpivirine
5. pregnant or breastfeeding women

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
H. pylori eradication rate of each group | UBT test 4 weeks after completion of eradication treatment
  H. pylori eradication rate of each group

CONTACTS AND LOCATIONS:
Locations (1):
- Incheon St. Mary's Hospital, Incheon, South Korea